CLINICAL TRIAL: NCT06486272
Title: The Financial Navigator Program - Optimizing Early Child Development by Facilitating Access to Financial Resources in the Neonatal Neurodevelopmental Follow-up Program
Brief Title: The Financial Navigator Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Edwin S.H. Leong Centre for Healthy Children (Unknown)
Responsible Party: Principal Investigator, Mathilda Vandenheuvel, Staff Pediatrician, Project Investigator, Associate Professor UofT, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000081699
Record Dates: First submitted 2024-06-19; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Financial Hardship
Keywords: Financial Services; Neonatal Neurodevelopment Follow-up Clinic
MeSH Terms: conditions — Financial Stress

STUDY DESIGN:
Intervention Model Description: Feasibility Pilot Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Financial Navigator Intervention (Experimental)
  Interventions: Other: Financial Navigator

INTERVENTIONS:
Other: Financial Navigator — Intervention: "Access to a Financial Navigator" We anticipate the Financial Navigator will meet at least 2 times and up to 2 additional visits, at a time convenient for the family. Examples of financial services that will likely be offered by the Financial Navigator are tax filing, applying for benefits and financial counseling. The program will be flexible and family centered. Families can choose if they would like to meet the Financial Navigator in person at the NNFU appointment, during another medical appointment, or at another time during a virtual visit. The Financial Navigator will be integrated into the existing SickKids Resource Navigation Service. At the 18-month NNFU visit the study will be completed.

SUMMARY:
Over one third of caregivers with a child admitted to the Hospital for Sick Children (SickKids) reported having difficulty making ends meet. The SickKids Medical-Financial Partnership (MFP) working group conducted in-depth interviews exploring financial needs and supports with selected caregivers in the Neonatal Neurodevelopmental Follow-up Program (NNFU). Results identified financial stress (including difficulties with employment, high cost of living, poverty, food insecurity, inaccessible supports, benefit time lines, costs of therapy) as a major theme. Caregivers generally supported the idea of hospital-based financial services. In this feasibility study we will trial a Financial Navigator Program in the NNFU.

DETAILED DESCRIPTION:
The objective of the current proposal will be to evaluate the feasibility of the Financial Navigator Program in the NNFU.

Research question: What is the feasibility of a Financial Navigator Program in the NNFU?

Setting: The NNFU program follows infants who had a Neonatal Intensive Care admission. Follow-up appointments are scheduled for when the infant is 4, 8, 12, 18 and 36 months of age. We will invite all families at their first appointment in the NNFU to participate in our study.

Study Procedure: Caregivers will be informed about the study at their child's first NNFU visit at 4 months. The clinical team will introduce the study and if interested, they will be approached by a Research Assistant (RA) to provide more details of the study. This can be in person at the clinic visit or in a follow-up phone call depended on families preference. If the caregiver provides consent, an appointment with the Financial Navigator will be arranged.

Intervention: "Access to a Financial Navigator" We anticipate the Financial Navigator will meet at least 2 times and up to 2 additional visits, at a time convenient for the family. Examples of financial services that will likely be offered by the Financial Navigator are tax filing, applying for benefits and financial counseling. The program will be flexible and family centered. Families can choose if they would like to meet the Financial Navigator in person at the NNFU appointment, during another medical appointment, or at another time during a virtual visit. The Financial Navigator will be integrated into the existing SickKids Resource Navigation Service. At the 18-month NNFU visit the study will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers with a child followed in the NNFU in SickKids will be invited to participate in our study.
* Caregiver needs to attend 4-month NNFU appointment.

Exclusion Criteria:

* There are no exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility; Measured with validated questionnaire including; Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), and Feasibility of Intervention Measure (FIM). | 14 months
  Validated Questionnaires (Weiner et al, 2017)
Demand | 14 months
  Demand will be evaluated by calculating the percentage of families that provided consent and the number of appointments per family with the Financial Navigator.

SECONDARY OUTCOMES:
Parenting Stress Index (PSI-Short Form) | 14 months
  Validated Questionnaire
Depression, Anxiety, Stress Scales (DASS) | 14 months
  Validated Questionnaire
Ages and Stages Questionnaire (ASQ) | 14 months
  ASQ 4 months and ASQ 18 month version
Economic outcomes | 14 months
  Standardized report: include tax filing, receipt of social assistance, Canada Tax Benefit and provincial tax benefit take up, parental leave benefits uptake, and reported uptake of other financial supports

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No